CLINICAL TRIAL: NCT03132597
Title: Impact of Teaching "Meditation Techniques" on the Mental Health and Quality of Life of Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 61240016.3.0000.5133
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-08

CONDITIONS: Stress; Anxiety; Depression; Quality of Life
Keywords: stress; anxiety; depression; quality of life; Mindfulness
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is an intervention protocol using a randomized controlled clinical trial with cross-over, in order to compare if the implementation of mindfulness for first year medical students will improve their mental health and quality of life in the short term (3 months).
  The intervention group will be exposed to mindfulness in the beginning of the medical course and will be compared to a control group, not exposed to mindfulness (exposed to theoretical classes) for 3 months. After that, the intervention group will receive theoretical classes and the control group will be exposed to the mindfulness techniques for 3 months (cross-over). Therefore, both groups will be exposed to mindfulness in the first year of undergraduation. Then, all first year medical students exposed to mindfulness will be compared to another class, which didn't have this mindfulness mandatory course in their formation. They will be compared after 6 months and after one-year of intervention (long-term effect).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Mindfulness exposure (Experimental): six weeks of 2 hours class of mindfulness training and orientations for home training at the beginning of the first semester
  Interventions: Behavioral: Mindfulness training
- Late Mindfulness exposure (Experimental): six weeks of 2 hours class of mindfulness training and orientations for home training at the second half of the first semester
  Interventions: Behavioral: Mindfulness training
- Control (not exposed) (No Intervention): Students not exposed to the mindfulness mandatory course (not exposed to the intervention)

INTERVENTIONS:
Behavioral: Mindfulness training — six weeks of 2 hours class of mindfulness training and orientations for home training
  Arms: Early Mindfulness exposure; Late Mindfulness exposure

SUMMARY:
Studies show a high number of medical students suffering from mental health problems. Although there are several studies investigating how these problems could impact students' life and performance, few studies have investigated interventions to minimize this distress. One of these interventions is the mindfulness meditation, that has already been extensively studied in the scientific literature showing promising results. Nevertheless, there are very few studies which investigated how mindfulness could be implemented as a mandatory course. The present study aims to investigate (1) how students exposed to mindfulness differ from students not exposed to this technique concerning their mental health and quality of life in a short and long term period. This is an intervention protocol using a randomized controlled clinical trial with cross-over, in order to compare if the implementation of mindfulness for first year medical students will improve their mental health and quality of life in the short term (3 months). The intervention group (group 1) will be exposed to mindfulness in the beginning of the medical course and will be compared to a control group (group 2), not exposed to mindfulness (exposed to theoretical classes) for 3 months. After that, the intervention group (group 1) will receive theoretical classes and the control group (group 2) will be exposed to the mindfulness techniques for 3 months (cross-over). Therefore, both groups will be exposed to mindfulness in the first year of undergraduation, however in different moments of the course. Then, these first year medical students (groups 1 and 2) will be compared to another class (group 3), which didn't have this mindfulness mandatory course in their formation. They will be compared after 6 months, 12 and 24 months of intervention (long-term effect).

DETAILED DESCRIPTION:
Studies show a high number of medical students suffering from mental health problems. Although there are several studies investigating how these problems could impact students' life and performance, few studies have investigated interventions to minimize this distress. One of these interventions is the mindfulness meditation, that has already been extensively studied in the scientific literature showing promising results. Nevertheless, there are very few studies which investigated how mindfulness could be implemented as a mandatory course. The present study aims to investigate how students exposed to mindfulness differ from students not exposed to this technique concerning their mental health and quality of life in a short and long term period.

Design:

This is an intervention protocol using a randomized controlled clinical trial with cross-over, in order to compare if the implementation of mindfulness for first year medical students will improve their mental health and quality of life in the short term (3 months).

The intervention group (group 1) will be exposed to mindfulness in the beginning of the medical course and will be compared to a control group (group 2), not exposed to mindfulness (exposed to theoretical classes) for 3 months. After that, the intervention group (group 1) will receive theoretical classes and the control group (group 2) will be exposed to the mindfulness techniques for 3 months (cross-over). Therefore, both groups (groups 1 and 2) will be exposed to mindfulness in the first year of undergraduation, however in different moments of the course. Then, all first year medical students exposed to mindfulness (groups 1 and 2) will be compared to another class, which didn't have this mindfulness mandatory course in their formation (group 3). They will be compared after 6 months and after one-year of intervention (long-term effect).

Interventions:

Mindfulness techniques will be delivered to students for a period of six weeks. In these six weeks the following techniques are presented and trained: body scan, mindful eating, breath meditation, listen mindfully, walking meditation, mountain meditation, compassion meditation, observation thoughts as just thoughts, awareness with listing of daily activities, mindful breath mini-breaks and some breath exercises.

Theoretical classes will provide tools in order to help students to deal with their medical school entrance, including how the medical school and the university works (library, evaluations, being a doctor, scholarships and student aid work, among others) and what students should know about their career as future physicians.

Procedures:

Students will answer the questionnaire in the following way:

* Intervention Group: before intervention (baseline), after intervention (3 months), after cross-over (6 months), 12 months and 24 months.
* Control Group: before intervention (baseline), before intervention (3 months), after intervention - cross over (6 months), 12 months and 24 months.
* Class not exposed to mindfulness mandatory course: 12 months and 24 months

Instruments:

The following instruments will be used:

* DASS-21: Depression, anxiety and stress scale
* Quality of Life: WHOQOL-Bref scale
* FFMQ: Five facet mindfulness questionnaire
* Sociodemographic data

Statistical analysis:

Students will be compared in the following way:

1. Students exposed to mindfulness versus students not exposed = short term period (3 months)
2. Students with an early exposition to mindfulness in the first year versus students with a later exposition = short term period (6 months)
3. Students exposed to a mandatory course on mindfulness versus students not exposed to this course = long term period (12 and 24 months)

ELIGIBILITY:
Inclusion Criteria:

* First year medical students who agree to participate in the study and are officially registered in the mindfulness course at the school of medicine - Federal University of Juiz de Fora, Brazil

Exclusion criteria:

* Students who refused to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assess emotional states of depression, anxiety and stress. | At 3 months
  DASS 21 questionnaire application
Assess emotional states of depression, anxiety and stress. | At 6 months
  DASS 21 questionnaire application
Assess emotional states of depression, anxiety and stress. | At 24 months
  DASS 21 questionnaire application

SECONDARY OUTCOMES:
Assess general facet of "quality of life" and "health" | At 3 months
  WHOQOL-BREF questionnaire application
Assess general facet of "quality of life" and "health" | At 6 months
  WHOQOL-BREF questionnaire application
Assess general facet of "quality of life" and "health" | At 24 months
  WHOQOL-BREF questionnaire application
Evaluation of empathy, spirituality openness and wellness | At 3 months
  ESWIM questionnaire application
Evaluation of empathy, spirituality openness and wellness | At 6 months
  ESWIM questionnaire application
Evaluation of empathy, spirituality openness and wellness | At 24 months
  ESWIM questionnaire application

CONTACTS AND LOCATIONS:
Overall Officials: Oscarina S Ezequiel, MD, PhD, Study Chair — Federal University of Juiz de Fora
Locations (1):
- Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbosa P, Raymond G, Zlotnick C, Wilk J, Toomey R 3rd, Mitchell J 3rd. Mindfulness-based stress reduction training is associated with greater empathy and reduced anxiety for graduate healthcare students. Educ Health (Abingdon). 2013 Jan-Apr;26(1):9-14. doi: 10.4103/1357-6283.112794. PMID 23823667
- [Background] de Vibe M, Solhaug I, Tyssen R, Friborg O, Rosenvinge JH, Sorlie T, Bjorndal A. Mindfulness training for stress management: a randomised controlled study of medical and psychology students. BMC Med Educ. 2013 Aug 13;13:107. doi: 10.1186/1472-6920-13-107. PMID 23941053
- [Background] Demarzo MM, Andreoni S, Sanches N, Perez S, Fortes S, Garcia-Campayo J. Mindfulness-based stress reduction (MBSR) in perceived stress and quality of life: an open, uncontrolled study in a Brazilian healthy sample. Explore (NY). 2014 Mar-Apr;10(2):118-20. doi: 10.1016/j.explore.2013.12.005. Epub 2013 Dec 18. No abstract available. PMID 24607079
- [Background] Dobkin PL, Hutchinson TA. Teaching mindfulness in medical school: where are we now and where are we going? Med Educ. 2013 Aug;47(8):768-79. doi: 10.1111/medu.12200. PMID 23837423
- [Background] Dyrbye LN, Thomas MR, Shanafelt TD. Systematic review of depression, anxiety, and other indicators of psychological distress among U.S. and Canadian medical students. Acad Med. 2006 Apr;81(4):354-73. doi: 10.1097/00001888-200604000-00009. PMID 16565188
- [Background] Ghodasara SL, Davidson MA, Reich MS, Savoie CV, Rodgers SM. Assessing student mental health at the Vanderbilt University School of Medicine. Acad Med. 2011 Jan;86(1):116-21. doi: 10.1097/ACM.0b013e3181ffb056. PMID 21099385
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Greeson JM, Toohey MJ, Pearce MJ. An adapted, four-week mind-body skills group for medical students: reducing stress, increasing mindfulness, and enhancing self-care. Explore (NY). 2015 May-Jun;11(3):186-92. doi: 10.1016/j.explore.2015.02.003. Epub 2015 Feb 16. PMID 25792145
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Background] Hojat M, Vergare MJ, Maxwell K, Brainard G, Herrine SK, Isenberg GA, Veloski J, Gonnella JS. The devil is in the third year: a longitudinal study of erosion of empathy in medical school. Acad Med. 2009 Sep;84(9):1182-91. doi: 10.1097/ACM.0b013e3181b17e55. PMID 19707055
- [Background] Jamali A, Tofangchiha S, Jamali R, Nedjat S, Jan D, Narimani A, Montazeri A. Medical students' health-related quality of life: roles of social and behavioural factors. Med Educ. 2013 Oct;47(10):1001-12. doi: 10.1111/medu.12247. PMID 24016170
- [Background] KABAT-ZINN, J. Full catastrophe living: Using the wisdom of your body and mind to face stress, pain and illness. New York: Delacorte, 1990.
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Kuhlmann SM, Burger A, Esser G, Hammerle F. A mindfulness-based stress prevention training for medical students (MediMind): study protocol for a randomized controlled trial. Trials. 2015 Feb 8;16:40. doi: 10.1186/s13063-014-0533-9. PMID 25887430
- [Background] Lamothe M, Rondeau E, Malboeuf-Hurtubise C, Duval M, Sultan S. Outcomes of MBSR or MBSR-based interventions in health care providers: A systematic review with a focus on empathy and emotional competencies. Complement Ther Med. 2016 Feb;24:19-28. doi: 10.1016/j.ctim.2015.11.001. Epub 2015 Nov 27. PMID 26860797
- [Background] Slavin SJ, Schindler DL, Chibnall JT. Medical student mental health 3.0: improving student wellness through curricular changes. Acad Med. 2014 Apr;89(4):573-7. doi: 10.1097/ACM.0000000000000166. PMID 24556765
- [Background] Tempski P, Bellodi PL, Paro HB, Enns SC, Martins MA, Schraiber LB. What do medical students think about their quality of life? A qualitative study. BMC Med Educ. 2012 Nov 5;12:106. doi: 10.1186/1472-6920-12-106. PMID 23126332
- [Background] van Dijk I, Lucassen PL, Speckens AE. Mindfulness training for medical students in their clinical clerkships: two cross-sectional studies exploring interest and participation. BMC Med Educ. 2015 Feb 25;15:24. doi: 10.1186/s12909-015-0302-9. PMID 25888726
- [Background] Warnecke E, Quinn S, Ogden K, Towle N, Nelson MR. A randomised controlled trial of the effects of mindfulness practice on medical student stress levels. Med Educ. 2011 Apr;45(4):381-8. doi: 10.1111/j.1365-2923.2010.03877.x. PMID 21401686
- [Background] Williams D, Tricomi G, Gupta J, Janise A. Efficacy of burnout interventions in the medical education pipeline. Acad Psychiatry. 2015 Feb;39(1):47-54. doi: 10.1007/s40596-014-0197-5. Epub 2014 Jul 18. PMID 25034955
- [Background] Moutinho IL, Maddalena NC, Roland RK, Lucchetti AL, Tibirica SH, Ezequiel OD, Lucchetti G. Depression, stress and anxiety in medical students: A cross-sectional comparison between students from different semesters. Rev Assoc Med Bras (1992). 2017 Jan 1;63(1):21-28. doi: 10.1590/1806-9282.63.01.21. PMID 28225885
- [Derived] Damiao Neto A, Lucchetti ALG, da Silva Ezequiel O, Lucchetti G. Effects of a Required Large-Group Mindfulness Meditation Course on First-Year Medical Students' Mental Health and Quality of Life: a Randomized Controlled Trial. J Gen Intern Med. 2020 Mar;35(3):672-678. doi: 10.1007/s11606-019-05284-0. Epub 2019 Aug 26. PMID 31452038